CLINICAL TRIAL: NCT05338957
Title: An Open-label, Multi-center, Phase I/II Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of MRG002 in Combination With HX008 in Patients With HER2-expressed Advanced Malignant Solid Tumors.
Brief Title: A Study of MRG002 in the Treatment of Patients With HER2-expressed Advanced Malignant Solid Tumors.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002/HX008-C001
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: MRG002; HX008; Antibody Drug Conjugate (ADC); HER2; PD-1; Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002+HX008 (Experimental): MRG002 will be administrated via intravenous infusion at 1.8，,2.2, or 2.6 mg/kg , (if appropriate) once on Day 1 of every 3 weeks (21-day cycle), up to 24 months.
  HX008 will be administrated via intravenous infusion at 3 mg/kg once on Day 1 of every 3 weeks (21-day- cycle), up to 24 months.
  Interventions: Drug: MRG002+HX008

INTERVENTIONS:
Drug: MRG002+HX008 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety and tolerability of MRG002 in combination with HX008 in patients with HER2-expressed advanced malignant solid tumors; and to , explore the maximum tolerated dose (MTD), and to determine the recommended phase II dose (RP2D) of combination therapy; , and to evaluate the preliminary efficacy, pharmacokinetics, and immunogenicity of combination therapy in the targeted study population.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form and follow the requirements specified in the protocol.
2. Aged 18 to 75 (including 18 and 75), both genders.
3. Life expectancy ≥ 12 weeks.
4. Patients with histopathological or cytological confirmed HER2-expressed advanced solid tumors, and with at least one measurable lesion according to the Response Criteria in Solid Tumors (RECIST v1.1).
5. The score of ECOG for performance status is 0 or 1.
6. The toxicity of previous anti-tumor treatment has recovered to ≤ Grade 1 as defined by NCI-CTCAEv5.0.
7. No severe cardiac dysfunction.
8. Organ functions must meet the basic requirements.
9. Cumulative dose of anthracycline ≤ 450 mg/m2 doxorubicin or its equivalent.

Exclusion Criteria:

1. Prior treatment with chemotherapy, biological therapy, immunotherapy, radiotherapy, investigational drugs, attenuated live vaccines, immunomodulators, CYP3A4 inhibitors/inducers, antibody-drug conjugates, etc.
2. Treatment with immune checkpoint inhibitors or tumor vaccines within 60 days prior to the first dose.
3. Treatment with systemic corticosteroids or other immunosuppressive drugs within 14 days prior to the first dose or during the study period.
4. History of severe cardiac disease.
5. Poorly controlled hypertension and hyperglycemia.
6. Presence of peripheral neuropathy ≥ Grade 2.
7. History of moderate or severe dyspnea at rest due to advanced malignant tumor or its complications or severe primary pulmonary disease, or current need of continuous oxygen therapy, or current interstitial lung disease or pneumonia.
8. Central nervous system metastasis.
9. Received major surgery within 4 weeks prior to the first dose without complete recovery.
10. History of hypersensitivity to any component of MRG002 or HX008 or known history of hypersensitivity of ≥ Grade 3 to macromolecular protein products/monoclonal antibodies.
11. Evidence of active infection.
12. History of primary immunodeficiency or autoimmune disease.
13. Female patients with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 6 months after the last dose of study treatment.
14. Previous history of other primary malignancies.
15. Other conditions inappropriate for participation in this study, as deemed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) in each dose group | Within 28 days after the first dose.
  DLT is defined as any of the treatment emergent adverse events (TEAE) as specified in the protocol that bear a definite, probable, or possible causal relationship to study drug administration within 28 days after the first dose.
Adverse events | After signing informed consent until 90 days after the last dose.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Recommended Phase II Dose (RP2D) | Baseline to study completion (up to 24 months)
  The dose level of MRG002 recommended for further clinical studies based on assessment of the safety, efficacy and PK data from this study.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (up to 24 months)
  ORR is defined as the proportion of subjects with CR and PR according to RECIST v1.1.
Duration of Response (DOR) | Baseline to study completion (up to 24 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and SD after treatment.
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Time to Response (TTR) | Baseline to study completion (up to 24 months)
  TTR is defined as the time from the start of treatment until the first occurrence of CR or PR by tumor assessment.
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.
PK parameters: concentration-time curve | Baseline to 90 days after the last dose.
  Plot of drug concentration changing with time after drug administration.
Immunogenicity (ADA) | Baseline to 90 days after the last dose.
  The proportion of patients with positive ADA results.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai Oriental Hospital
Locations (5):
- China (5):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No